CLINICAL TRIAL: NCT00569816
Title: A Comparison Between Continuous and Repetitive Sevoflurane Administration for Preconditioning During Coronary Artery Bypass Surgery
Brief Title: Continuous Versus Repetitive Sevoflurane Administration for Preconditioning
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Department of Anaesthesiology and Intensive Care Medicine (Ambiguous); Abbott (Industry)
Responsible Party: Prof. Dr. Jens Scholz, University Hospital Schleswig-Holstein, Campus Kiel, Department of Anaesthesiology and Intensive Care Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKSHCK-Anae07/06; ACA-GmbH-03-7
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2007-12-07 (Estimated); Status verified 2007-11

CONDITIONS: Myocardial Injury
Keywords: myocardial protection; pharmacological preconditioning; volatile anesthetics; myocardial injury following CABG surgery
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): Propofol as the primary anesthetic
  Interventions: Drug: Sevoflurane
- Group 2 (Experimental): Sevoflurane administered continuously after induction of anesthesia until initiation of cardiopulmonary bypass.
  Interventions: Drug: Sevoflurane
- Group 3 (Experimental): Sevoflurane administered repetitive up to 1 MAC from induction of anesthesia until initiation of cardiopulmonary bypass. Wash in and wash out performed twice.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — 1 MAC Sevoflurane will be given either continuously after induction of anesthesia until initiation of cardiopulmonary bypass or will be repetitively washed in and out twice before initiation of cardiopulmonary bypass.

SUMMARY:
Pharmacologic preconditioning by volatile anesthetics may depend on the mode of administration. The researchers hypothesize that a continuous administration in patients scheduled for CABG surgery prebypass will be less effective in terms of attenuating myocardial cell damage compared to a repetitive administration with a double wash in/wash out schedule. A control group will receive propofol as their primary anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Patients schedulded to undergo CABG surgery
* Age 18 to 80 years
* Ejection fraction > 40%

Exclusion Criteria:

* Emergency cases
* Diabetes
* Not able to give informed consent
* Ejection fraction < 40%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-01; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Myocardial cell damage as assessed by plasma levels of Troponin T | from induction of anesthesia until hospital discharge

SECONDARY OUTCOMES:
Length of stay on the ICU and in the hospital | from hospital admission until hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jens Scholz, MD, Principal Investigator — University Hospital Schleswig-Holstein, Campus Kiel, Department of Anaesthesiology and Intensive Care Medicine
Locations (1):
- University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Germany